CLINICAL TRIAL: NCT03295370
Title: Electrical Stimulation of Accessory Spinal Nerve in Cortical Activation, Muscular Perfusion and Autonomic Response in Healthy Subjects: a Randomized, Crossover, Sham Controlled Trial.
Brief Title: Electrical Stimulation of Accessory Spinal Nerve in Cortical Activation and Autonomic Response in Healthy Subjects
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Hospital de Clinicas de Porto Alegre (Other)
Responsible Party: Principal Investigator, Wolnei Caumo, Surgery Department Professor, School of Medicine UFRGS - MD. PhD., Hospital de Clinicas de Porto Alegre
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: 54489816.3.0000.5327
Record Dates: First submitted 2017-07-27; First posted 2017-09-27 (Actual); Last update posted 2018-01-05 (Actual); Status verified 2018-01

CONDITIONS: Pain
Keywords: Pain mechanisms; Cortical activation; fNIRS; Accessory spinal nerve; Autonomic response; Muscular perfusion
MeSH Terms: conditions — Pain | interventions — Electric Stimulation; Electroacupuncture

STUDY DESIGN:
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Active Group (Experimental): Needle electrical stimulation of accessory spinal nerve
  Interventions: Procedure: Electrical Stimulation
- Sham Group (Sham Comparator): Needle of accessory spinal nerve without electrical stimulation
  Interventions: Procedure: Electrical Stimulation

INTERVENTIONS:
Procedure: Electrical Stimulation — A needle is placed near accessory spinal nerve; electrical burst stimulation for 12 minutes, 10 Hz;
  Other Names: electroacupuncture

SUMMARY:
This randomized, crossover sham controlled trial with sham intended to study the effect of electrical stimulation on peripheral nerve (spinal accessory nerve) with acupuncture needle in healthy subjects aims to access the effect o electrical stimulation of accessory spinal nerve in cortical activation, muscular perfusion and autonomic response in healthy subjects.

Participants will be assessed through measure changes in cortical activation, local muscular peripheral perfusion and autonomic responses before and after intervention and intervention-sham, and crossed after a period of wash-out.

The design aims to contribute to assessment of one electroacupuncture's techniques by measuring some of the physiological effects caused by peripheral stimulation.

DETAILED DESCRIPTION:
In recent years, there are growing evidence that many diseases such as chronic pain and psychiatric disorders can be managed with non-pharmacological techniques. The possibility of inducing central neuroplastic responses through transcranial magnetic stimulation (TMS) and transcranial direct current stimulation (tDCS) has been widely studied, as well as peripheral stimulation techniques such electroacupuncture (EA) and intramuscular stimulation (IMS). However, there are few studies on physiological mechanisms, indications and limitations of each technique.

Thus, this randomized, crossover sham controlled trial, where sham intended to study the effect of electrical stimulation on peripheral nerve (spinal accessory nerve) with acupuncture needle in healthy subjects aims to access the effect o electrical stimulation of accessory spinal nerve in cortical activation, muscular perfusion and autonomic response in healthy subjects.

Participants will be assessed through measure changes in cortical activation, local muscular peripheral perfusion and autonomic responses before and after intervention and intervention-sham, and crossed after a period of wash-out.

The design aims to contribute to assessment of one electroacupuncture's techniques by measuring some of the physiological effects caused by peripheral stimulation.

ELIGIBILITY:
Inclusion Criteria:

* healthy male subjects
* right handed
* basic education

Exclusion Criteria:

* contraindication to infrared technology NIRS
* brain stimulator device
* drug and alcohol abuse
* chronic disease (any);
* chronic pain condition
* tobacco use
* psychiatric disorders
* Beck Depression Inventory higher then score 12
* psychotropic drugs
* use of pain-killers or anti-inflammatories 12h previous experiment

Ages: 18 Years to 55 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 14 (Actual)
Dates: Start 2017-06-13 (Actual); Primary Completion 2018-01-04 (Actual); Study Completion 2018-01-04 (Actual)

PRIMARY OUTCOMES:
Cortical Activation | 12 minutes
  The metabolic activation of motor cortex and dorsolateral prefrontal cortex , measured through infrared spectroscopy (fNIRS)

SECONDARY OUTCOMES:
Muscular perfusion | 12 minutes
  Muscular perfusion of trapezius muscle, peripherally measured through infrared spectroscopy (fNIRS)
Blood pressure | 20 minutes
  blood pressure measurement
Oxygen saturation | 20 minutes
  Oxygen measurement
Cardiac frequency | 20 minutes
  Cardiac frequency measurement

CONTACTS AND LOCATIONS:
Locations (1):
- Hospital de Clinicas e Porto Alegre (HCPA), Porto Alegre, Rio Grande do Sul, Brazil

IPD SHARING:
Plan to Share IPD: Undecided

REFERENCES:
- [Derived] Bandeira JS, Antunes LDC, Soldatelli MD, Sato JR, Fregni F, Caumo W. Functional Spectroscopy Mapping of Pain Processing Cortical Areas During Non-painful Peripheral Electrical Stimulation of the Accessory Spinal Nerve. Front Hum Neurosci. 2019 Jun 13;13:200. doi: 10.3389/fnhum.2019.00200. eCollection 2019. PMID 31263406